CLINICAL TRIAL: NCT03027518
Title: WILD 5 Wellness: A 30-Day Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beloit College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 302
Record Dates: First submitted 2017-01-17; First posted 2017-01-23 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Group 1 will be active in the WILD 5 Wellness program the first 30 days and inactive the 2nd 30 days.
  Interventions: Other: WILD 5 Wellness
- Group 2 (Other): Group 2 will be inactive in the WILD 5 Wellness program the first 30 days and active the 2nd 30 days.
  Interventions: Other: WILD 5 Wellness

INTERVENTIONS:
Other: WILD 5 Wellness — Participants will be asked to voluntarily engage in integrated, prescriptive, and trackable wellness interventions combining five wellness elements including exercise, mindfulness, sleep, social connectedness, and nutrition.

SUMMARY:
The purpose of this study is to explore the efficacy and feasibility of an integrated, prescriptive, and trackable wellness intervention combining five wellness elements including exercise, mindfulness, sleep, social connectedness, and nutrition in Beloit College students. This program is called "WILD 5 Wellness: A 30-Day Intervention". Results for this study will be quantified through the use of standardized self-report questionnaires administered prior to and after students complete the WILD 5 program (Group 1) or 30 days of inactive participation (Group 2), and again approximately 30 days later when the initially inactive group (Group 2) will have just completed their active participation in the WILD 5 program and the first WILD 5 group (Group 1) will be approximately 30 days out from completion of their WILD 5 active portion. Data will be collected to evaluate participants' adherence and response to each element of WILD 5, a 5-pronged 30-day wellness intervention. It is expected that this 30-day integrated, prescriptive, and trackable program will be found to be an efficacious wellness intervention for Beloit College students as compared to the control (inactive) group of students not participating in the Active program.

ELIGIBILITY:
Inclusion Criteria:

* Beloit College student enrolled in one or more of the following Spring 2017 academic courses:
* Anthropology 201 01 "Research Designs: Sophomore Seminar in Anthropology"
* Health and Society 240 B1 "Sophomore Seminar in Health and Society"
* Spanish 218 "Health and Culture in the Spanish-Speaking World"
* Biology 373 "Neuroscience Research"
* Biology 215 "Emerging Diseases"

Exclusion Criteria:

* Individuals who are <18 years old
* Individuals who are acutely suicidal and/or actively psychotic
* Individuals who are pregnant or plan to get pregnant during the next 60 days, or who are not registered in one of the courses listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
WILD 5 Wellness Scale (W5WS), Assessing Change | Day 0, Day 30, Day 60, Day 30 + 6 months (Group 1), Day 60 + 6 months (Group 2)
WILD 5 Wellness Elements (W5WE), Assessing Change | Day 0, Day 30, Day 60, Day 30 + 6 months (Group 1), Day 60 + 6 months (Group 2)
WILD 5 Wellness Effort Scale (W5WES), Assessing Change | Day 0, Day 30, Day 60, Day 30 + 6 months (Group 1), Day 60 + 6 months (Group 2)
WHO (World Health Organization) 5 Well-Being Index (1998 version), Assessing Change | Day 0, Day 30, Day 60, Day 30 + 6 months (Group 1), Day 60 + 6 months (Group 2)
Social Connectedness Scale (SCS), Assessing Change | Day 0, Day 30, Day 60, Day 30 + 6 months (Group 1), Day 60 + 6 months (Group 2)
Sleep Condition Indicator (SCI), Assessing Change | Day 0, Day 30, Day 60, Day 30 + 6 months (Group 1), Day 60 + 6 months (Group 2)
Sheehan Disability Scale (SDS), Assessing Change | Day 0, Day 30, Day 60, Day 30 + 6 months (Group 1), Day 60 + 6 months (Group 2)
Patient Health Questionnaire (PHQ-9), Assessing Change | Day 0, Day 30, Day 60, Day 30 + 6 months (Group 1), Day 60 + 6 months (Group 2)
Mindful Attention Awareness Scale (MAAS), Day to Day Experiences, Assessing Change | Day 0, Day 30, Day 60, Day 30 + 6 months (Group 1), Day 60 + 6 months (Group 2)
MIND ( Mediterranean-DASH Intervention for Neurodegenerative Delay)Diet, Assessing Change | Day 0, Day 30, Day 60, Day 30 + 6 months (Group 1), Day 60 + 6 months (Group 2)
Generalized Anxiety Disorder (GAD-7), Assessing Change | Day 0, Day 30, Day 60, Day 30 + 6 months (Group 1), Day 60 + 6 months (Group 2)
Eating and Appraisal Due to Emotions and Stress Questionnaire (EADES), Assessing Change | Day 0, Day 30, Day 60, Day 30 + 6 months (Group 1), Day 60 + 6 months (Group 2)
Cognitive and Physical Functioning Questionnaire (CPFQ), Assessing Change | Day 0, Day 30, Day 60, Day 30 + 6 months (Group 1), Day 60 + 6 months (Group 2)
Post Program Participant Questionnaire | The end of the 30 day active participation in WILD 5 Wellness for each group (1 and 2)

CONTACTS AND LOCATIONS:
Locations (1):
- Beloit College, Beloit, Wisconsin, United States